CLINICAL TRIAL: NCT02163018
Title: A First-in-human, Randomized, Double Blind, Placebo Controlled, Single-centre Study to Assess the Safety and Tolerability of HAL-MPE1 in Patients With Peanut Allergy
Brief Title: HAL-MPE1 First-in-human
Acronym: HAL-MPE1/0043
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HAL-MPE1/0043; 2013-004238-13 (EudraCT Number)
Record Dates: First submitted 2014-06-05; First posted 2014-06-13 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAL-MPE1 (Experimental): Subcutaneous administration of increasing doses of HAL-MPE1.
  Interventions: Drug: HAL-MPE1
- Placebo (Placebo Comparator): Subcutaneous administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HAL-MPE1 — Subcutaneous administration of increasing doses of HAL-MPE1
  Other Names: HAL-MPE1: modified peanut extract
  Arms: HAL-MPE1
Drug: Placebo — Subcutaneous administration of increasing doses of placebo
  Other Names: HAL-MPE1 placebo
  Arms: Placebo

SUMMARY:
Currently, there is no effective causal treatment for peanut allergy. A chemically modified, aluminium hydroxide adsorbed peanut extract (HAL-MPE1) for subcutaneous administration has been developed. Results from in vitro and in vivo preclinical studies demonstrate the immunotherapeutic potential of HAL-MPE1. Therefore, a phase I, single-centre clinical trial has been designed to assess the safety and tolerability of HAL-MPE1 in peanut allergic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female subjects aged 18-65 years.
3. A well-documented medical history of systemic reactions after ingestion of peanut
4. Positive food challenge at ≤1.5 gram peanut protein ingestion within the last 2 years
5. Positive serum specific anti-peanut and Ara h 2 Immunoglobulin E (IgE-test) (>0.7 kiloUnits(kU)/L) within the last 2 years
6. Forced expiratory volume at one second (FEV1)>70% of predicted value

Exclusion Criteria:

1. Subjects with a history of severe anaphylaxis to peanut with the following symptoms: hypotension, hypoxia, neurological compromise (collapse, loss of consciousness or incontinence) during challenge with peanuts.
2. Baseline serum tryptase level >20 µg/l
3. Known allergy or known hypersensitivity to (placebo) excipients
4. Participation in any interventional study aimed at desensitizing the peanut allergy in the past
5. Any specific immunotherapy (SCIT, SLIT or OIT) during the study period
6. Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
7. Significant active malignancies or any malignant disease within the past 5 years
8. Severe uncontrolled diseases that could increase the risk for patients participating in the study, including but not limited to: any severe or unstable lung diseases; endocrine diseases; clinically significant renal or hepatic diseases, or haematological disorders; or severe ongoing symptomatic allergic diseases
9. History of cardiovascular disease, uncontrolled hypertension or arrhythmias
10. Diseases with a contraindication for the use of adrenaline (e.g. hyperthyroidism, glaucoma)
11. Use of systemic steroids within 4 weeks before start of the study and during the study
12. Treatment with β-blockers/ACE inhibitors
13. Vaccination within one week before start of therapy or during study
14. Anti-IgE/anti-Tumor necrosis factor (TNF) therapy or any biologic immunomodulatory therapy within the 6 months prior to inclusion and during the study
15. Participation in a clinical study with a new investigational drug within the last 3 months or for a biological within the last 6 months prior to or during the study
16. Pregnancy (test performed at screening), lactation or inadequate contraceptive measures for women of child-bearing age (contraceptive measures considered adequate are: intrauterine devices, hormonal contraceptives, such as contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release)
17. Alcohol, drug or medication abuse within the past year
18. Any clinically significant abnormal laboratory parameter at screening
19. Lack or expected lack of cooperation or compliance
20. Severe psychiatric, psychological, or neurological disorders
21. Patients who are employees of the sponsor, institution or 1st grade relatives or partners of the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety of a SCIT-treatment with HAL-MPE1 in patients with peanut allergy. | up to 20 weeks
  * Occurrence of early and late local reactions
  * Occurrence of early and late systemic reactions
  * Occurrence of adverse events (clinically relevant abnormalities of the physical examination will be documented as adverse events)
  * Changes in laboratory values, vital signs, ECG and lung function.

SECONDARY OUTCOMES:
Change in serum levels of allergen specific immunoglobulins | before and after 15-20 weeks of treatment
Change in basophil histamine release test | before and after 15-20 weeks treatment
Change in titrated skin prick test | before and after 15-20 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bindslev-Jensen, Prof. Dr., Principal Investigator — Hudafdeling I og Allergicentret, Odense Universitetshospital
Locations (1):
- Carsten Bindslev-Jensen, Odense, Denmark